CLINICAL TRIAL: NCT01838018
Title: Brain Perfusion in Pantothenate Kinase-Associated Neurodegeneration (PKAN)
Status: Completed | Type: Observational
Sponsor: Susan J. Hayflick (Other)
Collaborators: Oregon Health and Science University (Other); Oregon Clinical and Translational Research Institute (Other)
Responsible Party: Sponsor-Investigator, Susan J. Hayflick, Professor & Chair, Molecular & Medical Genetics, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Other Study IDs: 8777
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Pantothenate Kinase-associated Neurodegeneration (PKAN)
Keywords: PKAN; brain iron; NBIA; neurodegeneration with brain iron accumulation; Hallervorden Spatz Syndrome
MeSH Terms: conditions — Pantothenate Kinase-Associated Neurodegeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PKAN: This group consists of individuals diagnosed with PKAN using a combination of MRI and PANK2 gene sequencing.
- Healthy volunteers: This is a control group of healthy volunteers, matched with the PKAN group for age and sex.

SUMMARY:
The purpose of this study is to learn whether blood flow in the brain is normal in people with pantothenate kinase-associated neurodegeneration (PKAN). Specifically, preliminary data suggest a region of the brain called the globus pallidus (GP), a key region affected by PKAN, may have reduced blood flow. Standard MRI and perfusion scanning techniques will be used to learn about cerebral blood flow in the globus pallidus and compare it to blood flow in other brain regions as well as to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PKAN confirmed by MRI and gene testing
* able to undergo MRI for approximately 1 hour without sedation

Exclusion Criteria:

* deep brain stimulators or other conditions that warrant avoidance of a strong magnetic field
* previous reaction to gadolinium (Gd) contrast agent
* acute or chronic kidney dysfunction
* pregnant and/or nursing at time of study

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The PKAN group consists of individuals in the United States diagnosed with PKAN.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
ASL-derived cerebral blood flow(CBF) | Single MRI
  The unit of analyses will be the subject and the primary comparison will be the globus pallidus CBF between PKAN and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Hayflick, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- See also: Related Info — http://www.ohsu.edu/xd/education/schools/school-of-medicine/departments/basic-science-departments/molecular-and-medical-genetics/people/primary-faculty/susan-hayflick.cfm